CLINICAL TRIAL: NCT02072018
Title: A Sequential, Randomized, Double-blind, Placebo-controlled, Prospective Study to Evaluate the Safety and Efficacy of the H-100 Treatment in Adult Male Volunteers With Peyronie's Disease
Brief Title: Peyronie's Disease Treatment Protocol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hybrid Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PDTP1
Record Dates: First submitted 2013-07-09; First posted 2014-02-26 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Peyronie's Disease
Keywords: Peyronie's; Peyronie's disease; Treatment; Clinical Study
MeSH Terms: conditions — Penile Induration | interventions — complement H100

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- H-100 (Active Comparator): H-100, gel, daily, 6 months
  Interventions: Drug: H-100
- Placebo (Placebo Comparator): Placebo gel, daily, three months then switch to H-100 for three months
  Interventions: Drug: H-100; Drug: Placebo

INTERVENTIONS:
Drug: H-100 — H-100 is a new compound to be applied to Peyronie's disease tissue with the intention of reducing disease symptoms.
Drug: Placebo — Placebo is an established, standard compound to be applied to Peyronie's disease tissue that will have no effect on disease symptoms.
  Arms: Placebo

SUMMARY:
Treatment of Peyronie's disease remains difficult. The purpose of this study is to test the safety and efficacy of a new compound to treat this disease.

ELIGIBILITY:
Inclusion Criteria:

1. Have symptom(s) of Peyronie's disease (pain, curvature or plaque)
2. Be judged to be in good health, based upon the results of a medical history, physical examination, and laboratory profile
3. Voluntarily sign and date an informed consent agreement approved by the Institutional Review Board/Independent Ethics Committee (IRB/IEC). The subject must also sign an authorization form to allow disclosure of his protected health information (PHI). The PHI authorization form and informed consent form may be an integrated form or may be separate forms depending on the institution
4. Be able to read, complete and understand the informed consent and various rating instruments in English

Exclusion Criteria:

1. Inability to understand study goals and risks
2. Inability to understand the informed consent
3. Inability to achieve erection with or without PDE5 inhibitor use adequate for penetration if penile curvature is not a limiting factor
4. Peyronie's disease symptoms greater than one year duration
5. Chordee in the presence or absence of hypospadias Thrombosis of the dorsal penile artery or vein Infiltration by a benign or malignant mass resulting in penile curvature Infiltration by an infectious agent, such as lymphogranuloma venereum Ventral curvature from any cause Presence of an active sexually transmitted disease Known active hepatitis B or C Known immune deficiency disease or be positive for human immunodeficiency virus (HIV)
6. Has previously undergone surgery for Peyronie's disease
7. Fails to have an erection which in the opinion of the investigator is sufficient to accurately measure the subject's penile deformity
8. Has an isolated hourglass deformity of the penis (curvature caused by a plaque that is noncontiguous with the hourglass deformity may be treated)
9. Has the plaque causing curvature of the penis located proximal to the base of the penis
10. Has previously received alternative medical therapies for Peyronie's disease administered by the intralesional route (including, but not limited to, steroids, verapamil, and the naturally occurring low molecular weight protein, interferon-α2b) within 3 months before the first dose of study drug or plans to use any of these medical therapies at any time during the study
11. Has received alternative medical therapies for Peyronie's disease administered by the oral (including, but not limited to, vitamin E [>500 U], potassium aminobenzoate [Potaba], tamoxifen, colchicine, pentoxifylline, over-the-counter erectile dysfunction medications, or steroidal anti-inflammatory drugs) or topical routes (including, but not limited to, verapamil applied as a cream) within 3 months before the first dose of study drug or plans to use any of these medical therapies at any time during the study
12. Has had extracorporeal shock wave therapy (ESWT) for the correction of Peyronie's disease within the 6- month period before screening or plans to have ESWT at any time during the study
13. Has used any mechanical type device for correction of Peyronie's disease within the 2-week period before screening or plans to use any these devices at any time during the study
14. Has used a mechanical device to induce a passive erection within the 2-week period before screening or plans to use any of these devices at any time during the study
15. Has significant erectile dysfunction that has failed to respond to oral treatment with phosphodiesterase type 5 (PDE5) inhibitors
16. Has uncontrolled hypertension, as determined by the investigator
17. Has a known recent history of stroke, bleeding, or other significant medical condition, which in the investigator's opinion would make the subject unsuitable for enrollment in the study
18. Is unwilling or unable to cooperate with the requirements of the study including completion of all scheduled study visits
19. Has received an investigational drug or treatment within 30 days before the first dose of study drug
20. Has a known systemic allergy to any H-100 component
21. Has received any collagenase treatments within 30 days of the first dose of study drug

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Safety measure | Up to six months
  Number of participants with adverse events. Continuous monitoring for adverse events. An adverse event is the development of an undesirable medical condition - e.g. symptoms or abnormal results of an investigation - or the deterioration of a pre-existing medical condition (not relevant in this study). Per the subject description, adverse events will be reported as: mild, moderate or severe.

SECONDARY OUTCOMES:
Efficacy measure | Up to three and six months (the Placebo group will change from Placebo to H-100 at the end of three months)
  Measure for change in pain, curvature, length, plaque hardness and plaque size. At the end of three months the Placebo group will change from Placebo to H-100 for the remaining three months. The H-100 group will receive H-100 for six months.
  Monitor for adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffry Twidwell, MD, Principal Investigator — North Memorial Medical Center
Locations (1):
- North Memorial Medical Center, Robbinsdale, Minnesota, United States